CLINICAL TRIAL: NCT06868212
Title: A US Phase 3b, Multi-center, Randomized, Double-blind, Double-Dummy Study to Evaluate Efficacy of Remibrutinib Compared to Dupilumab at Early Timepoints in Adults With Chronic Spontaneous Urticaria Inadequately Controlled by Second Generation H1-Antihistamines
Brief Title: A Study to Evaluate Efficacy of Remibrutinib Compared to Dupilumab at Early Timepoints in Adults With Chronic Spontaneous Urticaria Inadequately Controlled by Second Generation H1-antihistamines
Acronym: RECLAIM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CLOU064AUS02
Record Dates: First submitted 2025-03-06; First posted 2025-03-10 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Chronic Spontaneous Urticaria (CSU)
Keywords: BTK inhibitor; chronic spontaneous urticaria; Urticaria activity score; Hives severity score; Itch severity score
MeSH Terms: conditions — Chronic Urticaria | interventions — remibrutinib; dupilumab; Injections

STUDY DESIGN:
Intervention Model Description: Participants will be stratified based on prior exposure to anti-IgE biologics. Eligible participants will be randomized in a 1:1 ratio to receive remibrutinib or dupilumab and remibrutinib matching placebo or placebo solution for injection, both as an add-on treatment to once daily standard label dose of sgH1-AH background therapy, until the Week 12 visit.
  At the end of the 12-week double-blind treatment period, and in case remibrutinib is not commercially available, participants from both arms will be given the choice to roll over into an optional open label extension (OLE) period and receive remibrutinib (25 mg b.i.d. p.o.) for 12 weeks (up to Week 24).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment group 1: Remibrutinib + Placebo (Experimental): Remibrutinib tablet (25 mg b.i.d. p.o.) + placebo solution for injection in pre-filled syringe (2 s.c. injections at baseline and then 1 s.c. injection every other week [Weeks 2-10])
  Interventions: Drug: Remibrutinib; Drug: Placebo solution for injection
- Treatment group 2: Dupilumab + remibrutinib matching placebo (Active Comparator): Dupilumab pre-filled syringe (600 mg loading dose [2 x 300 mg dupilumab s.c. injection] at baseline visit followed by dupilumab 300 mg s.c. injection every other week [Weeks 2-10]) + remibrutinib matching placebo tablet (1 tablet b.i.d. p.o.)
  Interventions: Drug: Remibrutinib matching placebo; Drug: Dupilumab

INTERVENTIONS:
Drug: Remibrutinib — Film-coated tablet, oral administration, 25 mg b.i.d.
  Arms: Treatment group 1: Remibrutinib + Placebo
Drug: Remibrutinib matching placebo — Film-coated tablet, oral administration, b.i.d.
  Arms: Treatment group 2: Dupilumab + remibrutinib matching placebo
Drug: Dupilumab — Solution for injection in pre-filled syringe 600 mg loading dose followed by 300 mg dose every 2 weeks
  Arms: Treatment group 2: Dupilumab + remibrutinib matching placebo
Drug: Placebo solution for injection — Solution for injection in pre-filled syringe every 2 weeks
  Arms: Treatment group 1: Remibrutinib + Placebo

SUMMARY:
This is a US, multi-center, randomized, double-blind, double-dummy, Phase 3b study to evaluate efficacy of remibrutinib (25 mg twice daily [b.i.d.] by mouth [p.o.]) compared to dupilumab (600 mg loading dose administered subcutaneously (s.c.) followed by 300 mg every 2 weeks s.c.) at early timepoints (4 weeks and earlier), when administered as an add-on treatment to second generation H1-antihistamines (sgH1-AH) (standard label dose as background therapy) in adult US participants with moderate to severe chronic spontaneous urticaria (CSU) inadequately controlled by sgH1-AHs.

DETAILED DESCRIPTION:
This study consists of a screening period (up to 4 weeks), a core treatment period (12 weeks double-blind, double-dummy), an optional open-label extension [OLE] period, and safety follow-up period.

Screening period: participants will have a screening period of a minimum of 7 days up to a maximum of 28 days to establish eligibility for the study. Participants meeting all the inclusion criteria and none of the exclusion criteria will be eligible to participate in the study.

Core treatment period (double-blind, double-dummy): approximately, 400 participants diagnosed with CSU inadequately controlled by sgH1-AH will be randomized in this study. Participants will be stratified based on prior exposure to anti-IgE biologics.

Eligible participants will be randomized in a 1:1 ratio to receive remibrutinib and placebo solution for injection or dupilumab and remibrutinib matching placebo, both as an add-on treatment to once daily standard label dose of sgH1-AH background therapy, until the Week 12 visit.

Additionally, all participants will be on a stable, standard label dose of a sgH1-AH ("background therapy") throughout the entire core treatment period (starting a minimum of 7 days prior to randomization until the end of Week 12). To treat unbearable symptoms of CSU, participants will be allowed to add more of the same sgH1-AH on an as-needed basis ("rescue therapy"). The total maximum daily dose of sgH1-AH (background plus rescue) should not exceed 4 tablets/day (4-fold the standard label dose).

Optional open-label extension [OLE] period: At the end of the 12-week double-blind treatment period, and in case remibrutinib is not commercially available, participants from both arms will be given the choice to roll over into an optional OLE safety period and receive remibrutinib (25 mg b.i.d. p.o.) for 12 weeks (up to Week 24).

Safety follow-up period:

* For participants who do not enter the OLE period: there will be a safety follow-up for 12 weeks with safety follow-up phone calls at Week 16 and Week 24 (Week 24 will be end of study).
* For participants who enter the OLE period: there will be 2 options at the end of Week 24:
* If remibrutinib is commercially available: participants will discontinue study treatment, perform their EOT visit and receive a safety follow-up phone call 4 weeks after the last dose of remibrutinib (this will be the EOS).
* If remibrutinib is not commercially available, participants may continue on remibrutinib 25 mg b.i.d. until its commercial availability and return for site visits for safety follow up and treatment dispensation every 3 months. When remibrutinib becomes commercially available, the participant will be contacted for a site visit to complete the EOT visit and will receive a safety follow-up phone call 4 weeks after the last dose of remibrutinib (this will be the EOS).

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age at the time of signing the informed consent
* CSU duration for ≥ 6 months prior to screening (defined as the onset of CSU determined by the Investigator based on all available supporting documentation)
* Diagnosis of CSU inadequately controlled by sgH1-AH at the time of randomization, defined as:
* The presence of itch and hives for ≥ 6 consecutive weeks prior to screening despite the use of sgH1-AH during the 7 days prior to randomization (Day 1):
* UAS7 score (range, 0-42) ≥ 16, and
* ISS7 score (range, 0-21) ≥ 6, and
* HSS7 score (range, 0-21) ≥ 6
* Documentation of hives within 3 months before randomization (either at screening and/or at randomization); or documented in the participants medical history
* Willing and able to complete an Urticaria Patient Daily Diary (UPDD) for the duration of the study and adhere to the study protocol
* Participants must not have had more than one missing UPDD entry (either morning or evening) in the 7 days prior to randomization (Day 1)

Exclusion Criteria:

* Previous use of remibrutinib or other bruton's tyrosine kinase (BTK) inhibitors
* Previous use of dupilumab
* Evidence of clinically significant cardiovascular (such as but not limited to myocardial infarction, unstable ischemic heart disease, NYHA Class III/IV left ventricular failure, arrhythmia and uncontrolled hypertension within 12 months prior to Visit 1), neurological, psychiatric, pulmonary, renal, hepatic (past history or current), endocrine or metabolic disorder, or immunodeficiency that, in the investigator's opinion, would compromise the safety of the participant, interfere with the interpretation of the study results or otherwise preclude participation or protocol adherence of the participant.
* Evidence of hematological disorders (including coagulation disorders or significant bleeding risk)
* History or evidence of gastrointestinal disease (including gastrointestinal bleeding, e.g., in association with use of nonsteroidal anti-inflammatory drugs (NSAID), that was clinically relevant (e.g., where intervention was indicated or requiring hospitalization or blood transfusion)
* Requirement for anti-platelet medication, except for acetylsalicylic acid up to 100 mg/d or clopidogrel up to 75 mg/d. The use of dual anti-platelet therapy (e.g., acetylsalicylic acid + clopidogrel) is prohibited.
* Requirement for anticoagulant medication (for example, warfarin or Novel Oral Anti-Coagulants [NOAC])
* History or current hepatic disease including but not limited to acute or chronic hepatitis, cirrhosis or hepatic failure or hepatic parameters at screening: Aspartate Aminotransferase (AST)/ Alanine Aminotransferase (ALT) levels more than 1.5x ULN or International Normalized Ratio (INR) > 1.5 at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2027-02-22 (Estimated); Study Completion 2027-05-17 (Estimated)

PRIMARY OUTCOMES:
Absolute change from baseline in Weekly Urticaria Activity Score (UAS7) at Week 4 | Baseline, Week 4
  The UAS7 is the sum of the Weekly Hives Severity (HSS7) score and the Weekly Itch Severity (ISS7) score, and ranges from 0-42. Weekly scores (HSS7 and ISS7 scores) will be derived by adding up the average daily scores of the 7 days preceding the visit.

SECONDARY OUTCOMES:
Improvement of severity of hives, assessed as absolute change from baseline in HSS7 score at Week 4 | Baseline, Week 4
  The hives (wheals) severity score, defined by number of hives, will be recorded by the participant twice daily in their eCOA device, on a scale of 0 (none) to 3. A weekly score (HSS7) is derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score is therefore 0 - 21.
Improvement of severity of itch, assessed as absolute change from baseline in ISS7 score at Week 4 | Baseline, Week 4
  The severity of the itch will be recorded by the participant twice daily in their eCOA device, on a scale of 0 (none) to 3 (severe). A weekly score (ISS7) is derived by adding up the average daily scores of the 7 days preceding the visit. The possible range of the weekly score is therefore 0 - 21.
Improvement of UAS7, assessed as absolute change from baseline in UAS7 score at Week 1 | Baseline, Week 1
  The UAS7 is the sum of the Weekly Hives Severity (HSS7) score and the Weekly Itch Severity (ISS7) score, and ranges from 0-42. Weekly scores (HSS7 and ISS7 scores) will be derived by adding up the average daily scores of the 7 days preceding the visit.
Percentage of participants with UAS7 ≤ 6 at Week 4 | Week 4
  Percentage of participants who achieved UAS7 ≤ 6 at Week 4. The UAS7 is the sum of the Weekly Hives Severity (HSS7) score and the Weekly Itch Severity (ISS7) score, and ranges from 0-42. Weekly scores (HSS7 and ISS7 scores) will be derived by adding up the average daily scores of the 7 days preceding the visit.
Percentage of participants with UAS7=0 at Week 4 | Week 4
  Percentage of participants who achieved UAS7 = 0 at Week 4. The UAS7 is the sum of the Weekly Hives Severity (HSS7) score and the Weekly Itch Severity (ISS7) score, and ranges from 0-42. Weekly scores (HSS7 and ISS7 scores) will be derived by adding up the average daily scores of the 7 days preceding the visit.
Percentage of participants with UAS7 ≤ 6 at Week 2 | Week 2
  Percentage of participants who achieved UAS7 ≤ 6 at Week 2. The UAS7 is the sum of the Weekly Hives Severity (HSS7) score and the Weekly Itch Severity (ISS7) score, and ranges from 0-42. Weekly scores (HSS7 and ISS7 scores) will be derived by adding up the average daily scores of the 7 days preceding the visit.

CONTACTS AND LOCATIONS:
Locations (101):
- United States (101):
  - Allervie Clinical Research, Birmingham, Alabama
  - Cahaba Derm and skin hlth ctr 27, Birmingham, Alabama
  - Research Solutions of Arizona, Litchfield Park, Arizona
  - Peak Dermatology, Payson, Arizona
  - Premier Allergy Asthma And Immunology, Phoenix, Arizona
  - Avacare Center for Dermatology, Phoenix, Arizona
  - Orso Health, Scottsdale, Arizona
  - Acuro Research Inc, Little Rock, Arkansas
  - First OC Dermatology, Fountain Valley, California
  - Ctr for Dermatology Clinical Res, Fremont, California
  - Allergy and Asthma Specialists Group, Huntington Beach, California
  - Orso Health, Long Beach, California
  - Ark Clinical Research, Long Beach, California
  - California Allergy and Asthma Medical Group, Los Angeles, California
  - Dermatology Research Associates, Los Angeles, California
  - One Of A Kind Clinical Research, Napa, California
  - Empire Clinical Research, Pomona, California
  - Allergy and Asthma Consultants, Redwood City, California
  - Integrative Skin Science and Res, Sacramento, California
  - UC Davis Neuromuscular Research Center, Sacramento, California
  - Therapeutics Clinical Research, San Diego, California
  - Integrated Research of Inland Inc, Upland, California
  - Allergy and Asthma Clin Res Inc, Walnut Creek, California
  - Asthma and Allergy Associates P C, Colorado Springs, Colorado
  - UCONN Health Dermatology, Farmington, Connecticut
  - Howard University Hospital Division of Geriatrics, Washington D.C., District of Columbia
  - Florida Ctr Allergy Asthma Research, Aventura, Florida
  - Skin Care Research Inc, Boca Raton, Florida
  - Skin Care Research LLC, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - University of MiamiHealth System, Miami, Florida
  - FXM Clinical Res Miami LLC, Miami, Florida
  - Miami Dade Medical Research, Miami, Florida
  - Eminat Research Group, Miramar, Florida
  - Ziaderm Research LLC, North Miami Beach, Florida
  - AllerVie Health, Panama, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - Lenus Research and Med Group LLC, Sweetwater, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Asthma Allergy Immunology Clin Res, Tampa, Florida
  - Conquest Research, Winter Park, Florida
  - AllerVie Clin Res Columbus GA, Columbus, Georgia
  - Cleaver Medical Group, Cumming, Georgia
  - Southeast Dermatology Specialists, Douglasville, Georgia
  - Aeroallergy Research Laboratories, Savannah, Georgia
  - The Allergy Group-Meridian Clinic, Meridian, Idaho
  - Northshore University Health System, Glenview, Illinois
  - Midwest Allergy Sinus Asthma SC, Normal, Illinois
  - Clinical Res Ctr of S Illinois, O'Fallon, Illinois
  - Asthma and Allergy Center of Chicago S C, River Forest, Illinois
  - Deaconess Clin Allerg Res Inst, Evansville, Indiana
  - Southern IN Clinical Trials, New Albany, Indiana
  - Family Allergy And Asthma Rsch Inst, Louisville, Kentucky
  - Allergy and Asthma Specialist P S C, Owensboro, Kentucky
  - Ochsner Health Center, Baton Rouge, Louisiana
  - Chesapeake Clinical Research Inc, Baltimore, Maryland
  - AllerVie Clin Res Glenn Dale, Glenn Dale, Maryland
  - Boston Specialists LLC, Boston, Massachusetts
  - Derm Institute West Michigan PLLC, Caledonia, Michigan
  - Revival Research Institute, Troy, Michigan
  - Somerset Skin Centre, Troy, Michigan
  - Clinical Research Institute, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - The Clinical Research Center, St Louis, Missouri
  - Washington University, St Louis, Missouri
  - Las Vegas Dermatology, Las Vegas, Nevada
  - Hudson Essex Allergy-Circuit Clinical, Belleville, New Jersey
  - Circuit Clinical Mercer Algy Pulm, Hamilton, New Jersey
  - Allergy Asthma Assoc Monmouth, Little Silver, New Jersey
  - Circuit Clinical, Riverdale, New Jersey
  - Equity Medical, The Bronx, New York
  - UNC DermatologyandSkinCancer Ctr, Chapel Hill, North Carolina
  - Bernstein Clinical Research Center, Cincinnati, Ohio
  - CR Services Acquisition US, Columbus, Ohio
  - Optimed Research LLC, Columbus, Ohio
  - Wright State University, Fairborn, Ohio
  - Toledo Institute of Clinical Research, Toledo, Ohio
  - Unity Clinical Research, Oklahoma City, Oklahoma
  - Vital Prospects Clinical Research Institute, Tulsa, Oklahoma
  - Oregon Medical Research Center, Portland, Oregon
  - Oregon Health Sciences University, Portland, Oregon
  - Allergy and Clinical Immunology Associates, Pittsburgh, Pennsylvania
  - Tribe Clinical Research LLC, Greenville, South Carolina
  - Allergic Disease and Asthma Center, Greenville, South Carolina
  - Charleston ENT and Allergy, North Charleston, South Carolina
  - National Allergy and Asthma Research LLS, North Charleston, South Carolina
  - International Clinical Research Tennessee, LCC, Murfreesboro, Tennessee
  - Arlington Center for Dermatology, Arlington, Texas
  - Orion Clinical Research, Austin, Texas
  - Bellaire Dermatology Associates, Bellaire, Texas
  - Reveal Research Institute, Dallas, Texas
  - Pharma Research and Amp Consult, Dallas, Texas
  - Western Sky Medical Research, El Paso, Texas
  - Center for Clinical Studies, Houston, Texas
  - Sante Clinical Research, Kerrville, Texas
  - RFSA Dermatology, San Antonio, Texas
  - Andante Research, San Antonio, Texas
  - University Of Utah, Murray, Utah
  - Allergy Associates of Utah, Sandy City, Utah
  - Bellingham Asthma Allergy and Immunology, Bellingham, Washington

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations. This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com